CLINICAL TRIAL: NCT07339722
Title: A Phase 1, Randomized, Investigator- and Participant-Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Characterize the Safety, Tolerability, and Pharmacokinetics of LY4515100 in Healthy Participants
Brief Title: A Study of LY4515100 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27789; J6V-MC-OIAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY4515100 of Part A (SAD) (Experimental): Single-ascending doses of LY4515100 will be given orally
  Interventions: Drug: LY4515100 via SAD
- LY4515100 of Part B (MAD) (Experimental): Multiple-ascending doses of LY4515100 will be given orally
  Interventions: Drug: LY4515100 via MAD
- Placebo Part A (Placebo Comparator): Placebo will be given orally
  Interventions: Drug: LY4515100 via SAD
- Placebo Part B (Placebo Comparator): Placebo will be given orally
  Interventions: Drug: LY4515100 via MAD

INTERVENTIONS:
Drug: LY4515100 via SAD — given orally
  Arms: LY4515100 of Part A (SAD); Placebo Part A
Drug: LY4515100 via MAD — given orally
  Arms: LY4515100 of Part B (MAD); Placebo Part B

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY4515100 when given orally to healthy participants. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. The study will last up to 30 days and will include six overnight stays.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and cardiac monitoring.
* Have a body mass index within the range of 18.5 to 32.0 kilograms per square meter (kg/m^2) (inclusive).
* Individuals of childbearing potential (IOCBP) are excluded from this trial.
* Individuals not of childbearing potential (INOCBP) may participate in this trial.

Exclusion Criteria:

* Have donated 500 milliliters (mL) of blood within 30 days prior to dosing.
* Have participated within the last 30 days in a clinical study involving an investigational medicinal product. If the previous investigational product (IP) has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed.
* Participants with hemoglobin outside of the local laboratory normal reference range for age and sex, which is judged to be clinically significant by the investigator.
* Participants with an estimated glomerular filtration rate <90 mL/min/1.73 m2.
* Have a 12-lead Electrocardiogram (ECG) abnormality that, in the opinion of the investigator,
* increases the risks associated with participating in the study
* may confound ECG data analysis
* Have used or intend to use over-the-counter or prescription medication including dietary or herbal medications within 7 days, or 14 days if the medication is a potential enzyme inducer, or 5 half-lives (whichever is longer), prior to dosing.
* Smoke more than 10 cigarettes per day or the equivalent, including electronic cigarettes, and are unable to abide by investigative site smoking restrictions.
* Have an average weekly alcohol intake that exceeds 14 units per week (males 65 years of age or younger) and 7 units per week (females and males greater than 65 years of age, if applicable)
* Show evidence of
* Human immunodeficiency virus (HIV) infection and/or positive human HIV antigen and/or antibodies
* hepatitis C and/or positive hepatitis C antibody
* hepatitis B and/or positive hepatitis B surface antigen.
* Have liver disease.
* Any clinical condition or procedure (for example, gastrointestinal obstruction, gastric bypass, or cholecystectomy) that may affect the absorption, distribution, or excretion of the study drug and confound pharmacokinetics (PK) assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with one or more serious adverse event(s) (SAEs) of LY4515100 | Day 1 up to Day 30
  SAEs of LY4515100

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve (AUC) of LY4515100 | Day 1 through Day 11
  PK: AUC of LY4515100
PK: Maximum Observed Drug Concentration (Cmax) of LY4515100 | Time Frame: Day 1 through Day 11
  PK: Cmax of LY4515100
PK: Time of maximum observed drug concentration (tmax) of LY4515100 | Day 1 through Day 11
  PK: tmax of LY4515100

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-877-CTLILLY (1-877-285-4559) or, Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No